CLINICAL TRIAL: NCT00167804
Title: Comparing Virtual Reality Therapy to Usual Treatment for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3520P; NCT00223886 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Exposure Therapy; Post Traumatic Stress Disorder; Treatment Outcome; Veterans; Virtual Reality
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Virtual Reality Exposure Therapy

ARMS (1):
- 1 (Other): Present Centered Therapy focuses on the veterans problems in the here and now. It uses a problem solving approach and avoids discussion of war related traumatic events.
  Interventions: Behavioral: Virtual Reality Exposure

INTERVENTIONS:
Behavioral: Virtual Reality Exposure — VRE uses computer generated environments to conduct exposure therapy.

SUMMARY:
Combat related Posttraumatic Stress Disorder (PTSD) is the most common chronic psychiatric disorder in the veteran population. Unfortunately, outcome studies of VA PTSD programs have failed to show efficacy. VA PTSD patients have been significantly less responsive to conventional therapies than other PTSD populations. Virtual Reality based exposure therapy (VRE) allows patients to feel immersed in highly interactive computer-generated environments. Within these environments patients can be exposed to anxiety-provoking stimuli in a gradual and controlled manner so that they can become desensitized to these stimuli and, in the case of PTSD, the traumatic memories evoked by these stimuli. The advantages of VRE include less reliance on the patient's ability to visualize traumatic memories and making it more difficult for patients to avoid memories during exposure therapy. It is also safer and more convenient than in vivo exposure. In this study twenty Vietnam veterans are randomly assign to either VRE or to a Treatment as Usual (TAU) control condition. Treatment would consist of ten ninety-minute individual psychotherapy sessions for both groups. Assessments would occur at pre-treatment, immediate post-treatment and at six months post-treatment.

DETAILED DESCRIPTION:
Combat related Posttraumatic Stress Disorder (PTSD) is the most common chronic psychiatric disorder in the veteran population. PTSD is often disabling and is characterized by intrusive re-experiencing of traumatic memories, avoidance/numbing, and increased arousal. An estimated 830,000 veterans currently have chronic PTSD symptoms. The VA has set up 145 specialized PTSD programs. Unfortunately, outcome studies of VA PTSD programs have failed to show efficacy. VA PTSD patients have been significantly less responsive to conventional therapies than other PTSD populations including traditional Imaginal Exposure Therapy. Virtual Reality based exposure therapy (VRE) allows patients to feel immersed in highly interactive computer-generated environments. Within these environments patients can be exposed to anxiety-provoking stimuli in a gradual and controlled manner so that they can become desensitized to these stimuli and, in the case of PTSD, the traumatic memories evoked by these stimuli. VRE therapy produced significant and lasting reductions in PTSD symptoms with Vietnam veterans (N=14) in two open trials at the Atlanta VA. Two case studies of successful PTSD treatment (one at the Boston VA and the other of a 9/11 survivor) provide additional support for VRE. The advantages of VRE include less reliance on the patient's ability to visualize traumatic memories and making it more difficult for patients to avoid memories during exposure therapy. It is also safer and more convenient than in vivo exposure. The proposed study would randomly assign twenty Vietnam veterans to either VRE or to a Treatment as Usual (TAU) control condition. Treatment would consist of ten ninety-minute individual psychotherapy sessions for both groups. Assessments would occur at pre-treatment, immediate post-treatment and at six months post-treatment. VRE would use Virtual Vietnam computer generated environments to desensitize patients to one or two of their most traumatic combat related memories. VRE patients would wear a Head Mounted Display (HMD) that fits over their eyes and ears. While in the HMD patients look into a stereoscopic computer display and receive audio input through a set of headphones. Patients have reported a strong sense of being present in a Vietnam-like place when in these environments. The therapist is in constant contact with the patient through a microphone connected to the HMD. Patients recount their traumatic experiences while the therapist augments these descriptions with visual and auditory combat-related stimuli at the appropriate moments in time. The therapist can control, on a moment-by-moment basis, the type and intensity of the VR exposure. The goal is to provide the necessary level of stimuli to help the patient become engaged enough, long enough, to desensitize to a traumatic memory without becoming overwhelmed by either the external stimuli provided by the VR or the internal stimulus of the traumatic memory. In the TAU condition therapy will focus on "here-and-now" issues with a problem solving focus of the type that VA PTSD patients usually receive. The primary outcome measure will be the Clinician Administered PTSD Scale. An Independent Assessor who will be blind to patients' treatment conditions will conduct assessments. To insure patient safety, the Scale of Suicide Ideation will be administered in both conditions once a week. Patients will be paid $75 for each of the two post-treatment assessments. The hypotheses are: (1) VRE will produce significant reductions in PTSD symptoms; (2) VRE will be significantly more effective than TAU; (3) VRE symptom reduction will be maintained on six-month follow-up assessment. VRE may be a powerful new tool in the treatment of PTSD. Controlled studies, like the one proposed, are needed to explore its utility.

ELIGIBILITY:
Inclusion Criteria:

* Vietnam Veterans with combat related Posttraumatic Stress Disorder

Exclusion Criteria:

* Active Substance Abuse
* Psychosis
* Bipolar Disorder
* Dementia
* Significant Cognitive Impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | Pre Tx, Post TX and 6 months Post Tx

SECONDARY OUTCOMES:
Mississippi-R Scale | Pre Tx, Post TX and 6 months Post Tx

CONTACTS AND LOCATIONS:
Overall Officials: David Ready, PhD MS, Principal Investigator — VA Medical Center, Decatur
Locations (1):
- VA Medical Center, Decatur, Decatur, Georgia, United States